CLINICAL TRIAL: NCT05819684
Title: A Phase I Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of SHR-4602 in HER2 Expressing or Mutated Advanced Malignant Solid Tumor Subjects
Brief Title: A Study of SHR-4602 in Subjects With Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-4602-I-101
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: This is an open-label, three-part study to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of SHR-4602 and preliminary anti-tumor efficacy in HER2 expressing or mutated advanced malignant solid tumor subjects. Include three stages: dose escalation, PK expansion, and efficacy expansion.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: Dose escalation (Experimental)
  Interventions: Drug: SHR-4602 for injection
- Part 2: PK expansion (Experimental)
  Interventions: Drug: SHR-4602 for injection
- Part 3: efficacy expansion (Experimental)
  Interventions: Drug: SHR-4602 for injection

INTERVENTIONS:
Drug: SHR-4602 for injection — be administered via intravenous (IV) infusion

SUMMARY:
This is an open-label, three-part study to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of SHR-4602 and preliminary anti-tumor efficacy in HER2 expressing or mutated advanced malignant solid tumor subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced/unresectable or metastatic solid tumor with HER2 expression or mutation that is refractory to or intolerable with standard treatment, or for which no standard treatment is available;
2. At least one measurable lesion based on RECIST v1.1 criteria;
3. ECOG PS score: 0-1 points;
4. Expected survival period ≥ 3 months;
5. Adequate organ function;
6. Must take one medically approved contraceptive measure;
7. Patients voluntarily joined the study and signed informed consent.

Exclusion Criteria:

1. Patients with known CNS metastasis or hepatic encephalopathy;
2. Suffering from peripheral neuropathy;
3. History of clinically significant lung diseases (e.g., interstitial pneumonia, pneumonitis, pulmonary fibrosis, and severe radiation pneumonitis) or suspected to have these diseases by imaging at screening period;
4. Patients with any active, known or suspected autoimmune disorder;
5. With known severe allergic reactions to any other monoclonal antibodies;
6. Patients with symptomatic ascites or pleural effusion requiring paracentesis and drainage, or patients who have undergone ascites or pleural effusion drainage within 2 weeks before the first dose;
7. Patients with other malignancies currently or within the past 5 years;
8. Uncontrolled cardiac diseases or symptoms;
9. With known hereditary or acquired bleeding (e.g., coagulopathy) or a tendency to clot (e.g., hemophiliacs);
10. Patients with other potential factors that may affect the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From Day 1 to 90 days after last dose
Maximum tolerated dose (MTD) | From Day 1 to 21 days after first dose
Dose Limiting Toxicities (DLT) | From Day 1 to 21 days after first dose
Recommended Phase 2 dose (RP2D) | From Day 1 to 90 days after last dose

SECONDARY OUTCOMES:
PK parameters of SHR-4602 for Injection: Cmax | the date of first dose to 30 days after last dose
PK parameters of SHR-4602 for Injection: AUC0-t | the date of first dose to 30 days after last dose
PK parameters of SHR-4602 for Injection: Tmax | the date of first dose to 30 days after last dose
PK parameters of SHR-4602 for Injection: T1/2 | the date of first dose to 30 days after last dose
ADA | the date of first dose up to 90 days after last dose
  Anti-drug antibody, Immunogenicity of SHR-4602 for Injection
ORR | the date of first dose up to 90 days after last dose
  Objective Response Rate, Efficacy endpoints of SHR-4602 for Injection，As assessed by RECIST v1.1
DCR | the date of first dose up to 90 days after last dose
  Disease control rate, Efficacy endpoints of SHR-4602 for Injection，As assessed by RECIST v1.1
DOR | the date of first dose up to 90 days after last dose
  Duration of response, Efficacy endpoints of SHR-4602 for Injection，As assessed by RECIST v1.1
PFS | the date of first dose up to 90 days after last dose
  Progression Free Survival, Efficacy endpoints of SHR-4602 for Injection，As assessed by RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided